CLINICAL TRIAL: NCT04369924
Title: Improving Measurement-Based Care in Youth Mental Health: A Comparison of Unidimensional and Multidimensional Approaches
Brief Title: Personalized Assessment of Client Experiences
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Vanderbilt University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amanda Jensen-Doss, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190535; R34MH118316 (NIH)
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Mental Disorder in Adolescence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unidimensional Measurement-Based Care (Experimental): Youth and caregivers will complete a symptom rating scale every session. Clinicians will receive feedback reports summarizing these data, including alerts indicating if the youth is on track for positive treatment outcomes. These feedback reports will be used to support clinical decision-making.
  Interventions: Behavioral: Unidimensional Measurement-Based Care
- Multidimensional Measurement-Based Care (Experimental): Youth and caregivers will complete battery of questionnaires covering multiple process and outcome domains every session. Clinicians will receive feedback reports summarizing these data, including alerts indicating if the youth is on track for positive treatment outcomes. These feedback reports will be used to support clinical decision-making.
  Interventions: Behavioral: Multidimensional Measurement-Based Care

INTERVENTIONS:
Behavioral: Unidimensional Measurement-Based Care — Youth and caregivers will complete a symptom rating scale every session. Clinicians will receive feedback reports summarizing these data, including alerts indicating if the youth is on track for positive treatment outcomes. These feedback reports will be used to support clinical decision-making.
  Arms: Unidimensional Measurement-Based Care
Behavioral: Multidimensional Measurement-Based Care — Youth and caregivers will complete battery of questionnaires covering multiple process and outcome domains every session. Clinicians will receive feedback reports summarizing these data, including alerts indicating if the youth is on track for positive treatment outcomes. These feedback reports will be used to support clinical decision-making.
  Arms: Multidimensional Measurement-Based Care

SUMMARY:
The purpose of this study is to compare two clinical approaches to youth mental health care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female youth between the ages of 11-17 years receiving mental health services at the participating clinics.
2. The treating clinician is participating in the study and determines that Measurement-Based Care (MBC) is appropriate for the youth.
3. If the family consents to complete additional research measures, one parent and/or primary caregiver must be available and willing to participate in all study assessments.
4. Adolescent and at least one parent/guardian are able to complete all study procedures in English or Spanish.

Exclusion Criteria:

* no other exclusion criteria

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1261 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Douglas, Ph.D., Principal Investigator — Vanderbilt University; Amanda Jensen-Doss, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Health Connect America, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared via the National Institute of Mental Health Data Archive (NDA).
Time Frame: Data will be shared according to the NDA timelines.
Access Criteria: Data access will be according to the NDA guidelines.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All data reflect adolescent characteristics. Caregivers were not participants in the study.
Period: Overall Study
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Started | 637 | 624
Completed at Least One Measurement-based Care Measure | 411 | 370
Consented to Complete Additional Research Measures | 67 | 54
Completed (This was defined as completing at least two measurement-based care measures.) | 335 | 285
Not Completed | 302 | 339
Not completed — Lost to Follow-up | 302 | 339

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care | Total
Number analyzed (Participants) | 637 | 624 | 1261
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (2.1) | 13.9 (2.0) | 14.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 339 | 678
  Male | 298 | 285 | 583
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 18 | 34
  Not Hispanic or Latino | 521 | 494 | 1015
  Unknown or Not Reported | 100 | 112 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 62 | 105
  White | 466 | 422 | 888
  More than one race | 16 | 16 | 32
  Unknown or Not Reported | 111 | 124 | 235
The Ohio Scales Problem Severity Scale Youth Report [Mean (Standard Deviation); unit: scores on a scale] — A youth-report measure of youth symptoms ranging from 0 to 100, with higher scores indicating higher general mental health symptoms. Population: This measure was only administered to participants who consented to completing additional research measures.
  scores on a scale
    number analyzed (Participants) | 42 | 32 | 74
    (all) | 19.1 (16.0) | 20.6 (16.2) | 19.8 (16.0)
The Ohio Scales Problem Severity Scale Caregiver Report [Mean (Standard Deviation); unit: scores on a scale] — A caregiver-report measure of youth symptoms ranging from 0 to 100, with higher scores indicating higher general mental health symptoms. Population: This measure was only administered to participants who consented to completing additional research measures.
  scores on a scale
    number analyzed (Participants) | 43 | 32 | 75
    (all) | 19.9 (13.9) | 19.3 (14.4) | 19.6 (14.0)
The Ohio Scales Problem Functioning Scale Youth Report [Mean (Standard Deviation); unit: scores on a scale] — A youth-report measure of youth functioning in a variety of areas of daily living ranging from 0 to 80, with higher scores indicating better functioning. Population: This measure was only administered to participants who consented to completing additional research measures.
  scores on a scale
    number analyzed (Participants) | 41 | 31 | 72
    (all) | 55.1 (16.6) | 53.9 (15.4) | 54.6 (16.0)
The Ohio Scales Problem Functioning Scale Caregiver Report [Mean (Standard Deviation); unit: scores on a scale] — A caregiver-report measure of youth functioning in a variety of areas of daily living ranging from 0 to 80, with higher scores indicating better functioning. Population: This measure was only administered to participants who consented to completing additional research measures.
  scores on a scale
    number analyzed (Participants) | 42 | 31 | 73
    (all) | 49.3 (17.6) | 47.7 (20.1) | 48.6 (18.6)
Symptoms & Functioning Severity Scale- Youth Report [Mean (Standard Deviation); unit: scores on a scale] — A youth-report measure of youth mental health symptoms. Scores are reported as a total score, ranging from 33 to 86, with higher scores indicating higher symptoms. Population: Not all randomized participants went on to complete the measurement-based care measures.
  scores on a scale
    number analyzed (Participants) | 342 | 299 | 641
    (all) | 52.1 (10.0) | 50.9 (10.0) | 51.6 (10.0)
Symptoms & Functioning Severity Scale- Caregiver Report [Mean (Standard Deviation); unit: scores on a scale] — A caregiver-report measure of youth mental health symptoms. Scores are reported as a total score, ranging from 30 to 82, with higher scores indicating higher symptoms. Population: Not all youth who were randomized to condition had caregivers who participated in treatment. Not all youth who were randomized to condition had caregivers who completed measurement-based care measures.
  scores on a scale
    number analyzed (Participants) | 220 | 184 | 404
    (all) | 49.6 (9.2) | 50.0 (8.9) | 49.8 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in The Ohio Scales Problem Severity Scale Youth Report
Description: A youth-report measure of youth symptoms ranging from 0 to 100, with higher scores indicating higher general mental health symptoms.
Time Frame: baseline, 12 weeks
Population: This measure was only administered to participants who consented to completing additional research measures. Many of these were then lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 9 | 2
score on a scale | -4.4 (9.7) | 4.92 (9.3)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .25, ANOVA; F test for time by condition interaction = 1.49

2. Primary Outcome: Change in The Ohio Scales Problem Severity Scale Caregiver Report
Description: A caregiver-report measure of youth symptoms ranging from 0 to 100, with higher scores indicating higher general mental health symptoms.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 11 | 5
score on a scale | -2.2 (7.8) | 5.4 (9.9)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .12, ANOVA; F test for time by condition interaction = 2.80

3. Primary Outcome: Change in The Ohio Scales Problem Functioning Scale Youth Report
Description: A youth-report measure of youth functioning in a variety of areas of daily living ranging from 0 to 80, with higher scores indicating better functioning.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 8 | 2
score on a scale | 5.5 (15.6) | -4.5 (12.0)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .70, ANOVA; F test for time by condition interaction = .70

4. Primary Outcome: Change in The Ohio Scales Problem Functioning Scale Caregiver Report
Description: A caregiver-report measure of youth functioning in a variety of areas of daily living ranging from 0 to 80, with higher scores indicating better functioning.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 10 | 5
score on a scale | 2.4 (6.5) | -13.4 (25.3)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .07, ANOVA; F test for time by condition interaction = 3.67

5. Primary Outcome: Change in Symptoms & Functioning Severity Scale- Youth Report
Description: A youth-report measure of youth mental health symptoms. Scores are reported as a total score, ranging from 33 to 86, with higher scores indicating higher symptoms.
Time Frame: baseline, up to 18 months
Population: We analyzed youth who completed at least two sets of measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 326 | 220
score on a scale | -3.7 (0.6) | -3.3 (0.4)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .82, Mixed Models Analysis; Slope = .16

6. Primary Outcome: Change in Symptoms & Functioning Severity Scale- Caregiver Report
Description: A caregiver-report measure of youth mental health symptoms. Scores are reported as a total score, ranging from 30 to 82, with higher scores indicating higher symptoms.
Time Frame: baseline, up to 18 months
Population: We analyzed data from caregivers who completed at least two sets of measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
Number analyzed (Participants) | 220 | 184
score on a scale | -2.3 (0.4) | -2.6 (0.4)
Statistical Analysis 1: Comparison: Unidimensional Measurement-Based Care vs Multidimensional Measurement-Based Care; Test type: Superiority; p = .59, Mixed Models Analysis; Slope = -2.41

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Unidimensional Measurement-Based Care | Multidimensional Measurement-Based Care
All-Cause Mortality (participants affected / at risk) | 0/637 | 0/624
Serious Adverse Events (participants affected / at risk) | 0/637 | 0/624
Other Adverse Events (participants affected / at risk) | 0/637 | 0/624

LIMITATIONS AND CAVEATS:
The purpose of this trial was to pilot study procedures for a fully-powered trial. The procedures for recruiting and retaining research subsample participants were not successful, leading to a small number of participants with available data on the Ohio Scales outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04369924/Prot_SAP_000.pdf